CLINICAL TRIAL: NCT03825029
Title: Can the Difference Between the Operative and Radiographic Cup Inclination Angle Be Reduced by Applying a Pillow Between the Patient's Legs in Total Hip Arthroplasty Performed In The Lateral Decubitus Position?
Brief Title: Pillow Use During Total Hip Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20190058
Record Dates: First submitted 2019-01-29; First posted 2019-01-31 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Arthroplasty, Replacement, Hip; Hip Replacement, Total

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pillow Group (Experimental): There will be a pillow placed between the patients legs during their operation.
  Interventions: Procedure: Pillow
- Control Group (No Intervention): They will receive a normal total hip arthroplasty.

INTERVENTIONS:
Procedure: Pillow — A pillow to lessen the angle differences between hips so that the acetabular component can be placed in an optimal position.
  Arms: Pillow Group

SUMMARY:
The purpose of this study is to find out whether placing a pillow between the legs during hip surgery will result in a better aligned hip replacement.

DETAILED DESCRIPTION:
During hip replacement surgery the cup is placed on specific planned angles. Cup placement has an effect on the patients' pain-free range of movement, dislocation rates and satisfaction. However, the angles of the cup orientation (i.e. the tilt and rotation), which are preoperatively planned and postoperatively measured on radiographs, have a high variability even when an experienced surgeon is performing the surgery. One of the reasons this occurs is because the operated leg can move the pelvis to a different position in the time between set-up and actual implantation which may lead to the cup being placed in a non-optimal position. This study aims to see if the difference between planned and achieved cup angles and pelvic movement can be lessened by putting a pillow in between the legs to keep it in a stable horizontal position.

ELIGIBILITY:
Inclusion Criteria:

* Patient awaiting primary total hip arthroplasty using a posterior approach in a lateral decubitus position
* Patients capable of reading, understanding, and willing to sign the informed consent form

Exclusion Criteria:

* Total hip arthroplasty not using a posterior approach in a lateral decubitus position
* Prior hip osteotomy or fracture osteosynthesis on the index hip

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-07-22 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Change in radiographic cup inclination angle | Intra-operatively and post-operatively (within one month after the surgery)
  The difference between the operative and postoperative radiographic cup inclination angle

CONTACTS AND LOCATIONS:
Overall Officials: George Grammatopoulos, MBBS BSc FRCS DPhil, Principal Investigator — The Ottawa Hospital Research Institute
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

REFERENCES:
- [Background] Ozaki Y, Baba T, Homma Y, Ochi H, Watari T, Banno S, Matsumoto M, Kaneko K. Posterior versus direct anterior approach in total hip arthroplasty: difference in patient-reported outcomes measured with the Forgotten Joint Score-12. SICOT J. 2018;4:54. doi: 10.1051/sicotj/2018051. Epub 2016 Nov 27. PMID 30480545
- [Background] Kennedy JG, Rogers WB, Soffe KE, Sullivan RJ, Griffen DG, Sheehan LJ. Effect of acetabular component orientation on recurrent dislocation, pelvic osteolysis, polyethylene wear, and component migration. J Arthroplasty. 1998 Aug;13(5):530-4. doi: 10.1016/s0883-5403(98)90052-3. PMID 9726318
- [Background] D'Lima DD, Urquhart AG, Buehler KO, Walker RH, Colwell CW Jr. The effect of the orientation of the acetabular and femoral components on the range of motion of the hip at different head-neck ratios. J Bone Joint Surg Am. 2000 Mar;82(3):315-21. doi: 10.2106/00004623-200003000-00003. PMID 10724224
- [Background] Grammatopoulos G, Thomas GE, Pandit H, Beard DJ, Gill HS, Murray DW. The effect of orientation of the acetabular component on outcome following total hip arthroplasty with small diameter hard-on-soft bearings. Bone Joint J. 2015 Feb;97-B(2):164-72. doi: 10.1302/0301-620X.97B2.34294. PMID 25628277
- [Background] Widmer KH. [Impingement Free Motion in Total Hip Arthroplasty - How Can We Implement It?]. Z Orthop Unfall. 2016 Aug;154(4):392-7. doi: 10.1055/s-0042-108065. Epub 2016 Jun 23. German. PMID 27336842
- [Background] Fujishiro T, Hiranaka T, Hashimoto S, Hayashi S, Kurosaka M, Kanno T, Masuda T. The effect of acetabular and femoral component version on dislocation in primary total hip arthroplasty. Int Orthop. 2016 Apr;40(4):697-702. doi: 10.1007/s00264-015-2924-2. Epub 2015 Jul 23. PMID 26202021
- [Background] Grammatopoulos G, Pandit HG, da Assuncao R, Taylor A, McLardy-Smith P, De Smet KA, Murray DW, Gill HS. Pelvic position and movement during hip replacement. Bone Joint J. 2014 Jul;96-B(7):876-83. doi: 10.1302/0301-620X.96B7.32107. PMID 24986939
- [Background] Meermans G, Goetheer-Smits I, Lim RF, Van Doorn WJ, Kats J. The difference between the radiographic and the operative angle of inclination of the acetabular component in total hip arthroplasty: use of a digital protractor and the circumference of the hip to improve orientation. Bone Joint J. 2015 May;97-B(5):603-10. doi: 10.1302/0301-620X.97B5.34781. PMID 25922452
- [Background] Wright JG. Small Simple Trials: A Strategy for Orthopaedic Randomized Trials. J Bone Joint Surg Am. 2018 Jul 18;100(14):e95. doi: 10.2106/JBJS.17.01107. No abstract available. PMID 30020133
- [Background] Langton DJ, Sprowson AP, Mahadeva D, Bhatnagar S, Holland JP, Nargol AV. Cup anteversion in hip resurfacing: validation of EBRA and the presentation of a simple clinical grading system. J Arthroplasty. 2010 Jun;25(4):607-13. doi: 10.1016/j.arth.2009.08.020. Epub 2009 Dec 21. PMID 20022454